CLINICAL TRIAL: NCT03355794
Title: A Phase I Study of Ribociclib and Everolimus Following Radiation Therapy in Children With Newly Diagnosed Non-biopsied Diffuse Pontine Gliomas (DIPG) and RB+ Biopsied DIPG and High Grade Gliomas (HGG)
Brief Title: A Study of Ribociclib and Everolimus Following Radiation Therapy in Children With Newly Diagnosed Non-biopsied Diffuse Pontine Gliomas (DIPG) and RB+ Biopsied DIPG and High Grade Gliomas (HGG)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CONNECT1701_LEE/RAD17T-MD-1604
Record Dates: First submitted 2017-11-22; First posted 2017-11-28 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Diffuse Intrinsic Pontine Glioma; Malignant Glioma of Brain; High Grade Glioma; Bithalamic High Grade Glioma; Brainstem Glioma; Glioblastoma; Anaplastic Astrocytoma
Keywords: DIPG; High Grade Glioma; ribociclib; everolimus
MeSH Terms: conditions — Diffuse Intrinsic Pontine Glioma; Glioma; Glioblastoma; Astrocytoma | interventions — ribociclib; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose level 1 (starting dose level) (participants </= 21yrs) (Experimental): Ribociclib administered orally; daily on days 1-21 each 28 day cycle; dose calculation age dependent (>21 yrs of age 300mg daily (DIPG only); </=21 yrs of age 120 mg/m2/day) Everolimus administered orally; daily on days 1 - 28 each 28 day cycle; dose calculation age dependent (>21yrs 2.5mg/day (DIPG only); </=21yr 1.2 mg/m2/day) BSA >/=0.75m2
  Interventions: Drug: ribociclib; Drug: Everolimus
- Dose level 2 (participants </= 21yrs) (Experimental): Ribociclib administered orally; daily on days 1-21 each 28 day cycle; 170 mg/m2/day Everolimus administered orally; daily on days 1 - 28 each 28 day cycle; 1.2 mg/m2/day BSA >/=0.45m2
  Interventions: Drug: ribociclib; Drug: Everolimus
- Dose level 3 (participants </= 21yrs) (Experimental): Ribociclib administered orally; daily on days 1-21 each 28 day cycle; 170 mg/m2/day Everolimus administered orally; daily on days 1 - 28 each 28 day cycle; 1.5 mg/m2/day BSA >/=0.45m2
  Interventions: Drug: ribociclib; Drug: Everolimus
- Dose level 1 (DIPG participants > 21yrs) (Experimental): Ribociclib administered orally; daily on days 1-21 each 28 day cycle; 300mg daily Everolimus administered orally; daily on days 1 - 28 each 28 day cycle; 2.5mg/day
  Interventions: Drug: ribociclib; Drug: Everolimus

INTERVENTIONS:
Drug: ribociclib — Oral capsule or liquid formula
  Other Names: Kisqali
Drug: Everolimus — Oral tablets or dispersible tablets
  Other Names: Afinitor

SUMMARY:
In this research study, we want to learn about the safety of the study drugs, ribociclib and everolimus, when given together at different doses after radiation therapy. We also want to learn about the effects, if any, these drugs have on children and young adults with brain tumors.

We are asking people to be in this research study who have been diagnosed with a high grade glioma, their tumor has been screened for the Rb1 protein, and they have recently finished radiation therapy. If a patient has DIPG or a Bi-thalamic high grade glioma, they do not need to have the tumor tissue screened for the Rb1 protein, but do need to have finished radiation therapy.

Tumor cells grow and divide quickly. In normal cells, there are proteins that control how fast cells grow but in cancer cells these proteins no longer work correctly making tumor cells grow quickly. Both study drugs work in different ways to slow down the growth of tumor cells. The researchers think that if the study drugs are given together soon after radiation therapy, it may help improve the effect of the radiation in stopping or slowing down tumor growth.

The study drugs, ribociclib and everolimus, have been approved by the United States Food and Drug Administration (FDA). Ribociclib is approved to treat adults with breast cancer and everolimus is approved for use in adults and children who have other types of cancers. The combination of ribociclib and everolimus has not been tested in children or in people with brain tumors and is considered investigational.

The goals of this study are:

* Find the safest dose of ribociclib and everolimus that can be given together after radiation.
* Learn the side effects (both good and bad) the study drugs have on the body and tumor.
* Measure the levels of study drug in the blood over time.
* Study the changes in the endocrine system that may be caused by the tumor, surgery or radiation.

DETAILED DESCRIPTION:
This is a phase I study to determine: 1) the MTD and/or the recommended phase II dose (RP2D) of ribociclib and everolimus which can be safely administered during maintenance therapy for up to 24 courses following completion of radiation therapy with newly diagnosed non-biopsied DIPG and RB+ biopsied DIPG and HGG, 2) characterization of the pharmacokinetic profile of ribociclib and everolimus as combination maintenance therapy following completion of radiation therapy with newly diagnosed non-biopsied DIPG and RB+ biopsied DIPG and HGG.

Patients with RB+ tumors and non-biopsied DIPG will receive standard radiation therapy prior to enrollment followed by ribociclib and everolimus as maintenance therapy. Upon completion of radiation therapy, a 2 - 4 week break will occur and then ribociclib will be given orally daily for 21 days followed by a 7 day break every 28 days at 70% of the adult RP2D (300 mg) in combination with everolimus at 80% of the adult RP2D (2.5 mg) given orally once daily continuously for up to 24 courses. One course is equivalent to 28 days. Due to dosing concerns with the limited dosing capsules (50 mg and 200 mg are only available), dose escalations will have BSA restrictions to accommodate for variations from target doses and BSA adjusted actual dose. Two intra-patient dose-de-escalations will be allowed if dose limiting toxicities arise and may continue study treatment for up to 24 courses in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Age Patients must be ≥ 12 months of age and ≤ 30 years of age at the time of study entry for patients diagnosed with DIPG.

Patients must be ≥ 12 months of age and ≤ 21 years of age at the time of study entry for patients diagnosed with HGG.

* BSA restrictions for patients ≤ 21 years of age at the time of study entry

  * Patients enrolled on dose level -1 must have BSA≥0.55m2
  * Patients enrolled on dose level 0* must have BSA≥0.75m2
  * Patients enrolled on dose level 0 must have BSA≥0.55m2
  * Patients enrolled on dose level 1 must have BSA≥0.75m2
  * Patients enrolled on dose level 2 and 3 must have BSA≥ 0.45m2
* RB status Screening for RB applies to all patients with pre-trial tumor tissue except for patients diagnosed with DIPG and bi-thalamic tumors who do not have available tissue.

RB testing must be evaluated centrally at CCHMC prior to enrollment or report from CLIA certified lab must be reviewed centrally at CCHMC.

* Tumor

Diffuse Intrinsic Pontine Glioma (DIPG):

Patients with newly diagnosed diffuse intrinsic pontine gliomas (DIPGs), defined on neuroimaging as tumors with a pontine epicenter and diffuse intrinsic involvement of the pons, are eligible without histologic confirmation.

Patients with brainstem tumors that do not meet these criteria or not considered to be typical intrinsic pontine gliomas will only be eligible if the tumors are biopsied and proven to have + RB and be the following according to the 2016 World Health Organization Classification of Tumors of the Central Nervous System proved to be high grade gliomas (such as anaplastic astrocytoma, glioblastoma, H3K27-mutant diffuse midline glioma or diffuse astrocytoma) Or histologically-confirmed malignant glioma WHO II-IV "other than above".

Note: Patients with juvenile pilocytic astrocytoma, pilomyxoid astrocytoma, pleomorphic xanthoastrocytoma with or without anaplasia, gangliogliomas, or other mixed gliomas without anaplasia are not eligible.

Patients with diffuse intrinsic brain stem glioma (DIPG) can be enrolled without the need for available tumor tissue for RB protein status confirmation. If DIPG or bi-thalamic patients have been biopsied and if available tissue, RB status will be tested. These must be RB+ to be eligible for enrollment.

Bi-thalamic tumors, biopsied and noted to have intact RB are eligible. Bi-thalamic tumors that are not biopsied will be eligible to enroll on the DIPG non-biopsied arm. 107

High-grade Glioma (HGG):

Patients with newly-diagnosed non-brainstem high-grade glioma (HGG) are eligible. Patients must have had histologically verified high-grade glioma such as anaplastic astrocytoma, glioblastoma, H3 K27 mutant diffuse midline glioma etc. Or histologically-confirmed non-brain stem malignant high grade glioma WHO III-IV "other than above".

AND RB+ noted on immunohistochemistry.

Patients with primary spinal cord tumors are eligible. Patients with multi-focal disease within the cerebrum are eligible.

Patients with a diagnosis of oligodendroglioma or oligoastrocytoma are not eligible.

* MRI of spine must be performed prior to enrollment if the treating physician suspects disseminated disease as a baseline evaluation. If leptomeningeal disease develops post radiation therapy and prior to enrollment, patients may be considered eligible if craniospinal irradiation was not received prior to enrollment.
* Performance Status Karnofsky ≥ 50% for patients >16 years of age or Lansky ≥50 for patients >16 years of age. Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
* Prior Therapy Patients must have not received any prior therapy other than surgery, radiation (focal to disease) and/or steroids (dexamethasone with goal to wean dexamethasone throughout protocol therapy).
* Radiation therapy requirements

  * Patients diagnosed with DIPG: any variances in the radiotherapy dose within 10% of the current standard dose (54 Gy) will be discussed with the Sponsor-Investigator to confirm eligibility prior to study enrollment.
  * Patients diagnosed with HGG: any variances in the radiotherapy dose within 10% of the current standard dose (59.4 Gy) will be discussed with the Sponsor-Investigator to confirm eligibility prior to study enrollment.
  * Patients diagnosed with primary spinal tumors any variances in the radiotherapy dose within 10% of the current standard dose (54 Gy) will be discussed with the Sponsor-Investigator to confirm eligibility prior to study enrollment.
  * Timing of Radiation Radiation therapy must have begun no later than 30 days after the date of radiographic diagnosis or definitive surgery, whichever is the later date.
* Organ Function Patients must have normal organ and marrow function documented within 7 days of study enrollment
* All patients must have recovered from all acute RT-related toxicities to ≤ grade 2 prior to initiating the use of ribociclib and everolimus.
* Pregnancy Status Female patients of childbearing potential, must not be pregnant or breast-feeding. Female patients of childbearing potential must have a negative serum or urine pregnancy test.
* Pregnancy Prevention Women of child-bearing potential are defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception throughout the study and for 8 weeks after study drug discontinuation.
* Female patients with infants must agree not to breastfeed their infants while on this study.
* Informed Consent Signed informed consent according to institutional guidelines must be obtained. Assent, when appropriate, will be obtained according to institutional guidelines.

Exclusion Criteria:

* Concurrent Illness Patients with any clinically significant unrelated systemic illness (serious infections or significant cardiac, pulmonary, hepatic or other organ dysfunction) that would compromise the patient's ability to tolerate protocol therapy or would likely interfere with the study procedures or results.
* Inability to Participate Patients with inability to return for follow-up visits or obtain follow-up studies required to assess toxicity to therapy.
* Received a radiosensitizer, craniospinal irradiation therapy, investigational agent or any additional adjuvant therapy during radiation therapy.
* Received prior therapy with CDK4/6 inhibitor and/or mTOR inhibitor.
* Seizures Patients who are currently receiving enzyme inducing anti-epileptic drugs that are known strong inducers or inhibitors of CYP3A4/5 (EIAEDs). Patients with a history of seizures and maintained on an anti-epileptic drug that is not a strong inducers or inhibitor of CYP3A4/5 are eligible.
* Patient has a known hypersensitivity to ribociclib or any of its excipients as described below:

  * The capsules contain only the drug substance without any excipients.
  * The film-coated tablets consist of drug substance and compendial quality colloidal silicon dioxide, crospovidone, hydroxypropylcellulose, magnesium stearate and microcrystalline cellulose. The film-coating is a mix of compendial quality iron oxides, lecithin, polyvinyl alcohol, talc, titanium dioxide, and xanthan gum. Patients allergic to peanut and soy are not permiteed to take the film-coated tablet formulation.
  * The oral solution consists of ribociclib succinate in water with an orange flavoring agent and common excipients such as preservatives, sweetener and pH modifier
* Clinically significant active cardiac disease, uncontrolled heart disease and/or history of cardiac dysfunction including any of the following;

  * History of acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass grafting, coronary angioplasty, or stenting) or symptomatic pericarditis within 12 months prior to screening
  * History of documented congestive heart failure (New York Heart Association functional classification III-IV)
  * Documented cardiomyopathy
  * Patient has a Left Ventricular Ejection Fraction (LVEF) <50% as determined by Multiple Gated acquisition (MUGA) scan or echocardiogram (ECHO) at screening
  * History of any cardiac arrhythmias, e.g., ventricular, supraventricular, nodal arrhythmias, or conduction abnormality within 12 months of screening
  * Long QT syndrome or known family history of idiopathic sudden death or congenital long QT syndrome, or any of the following:

    * Risk factors for Torsades de Pointe (TdP) including uncorrected hypokalemia or hypomagnesemia, history of cardiac failure, or history of clinically significant/symptomatic bradycardia.
    * Concomitant use of medication(s) with a known risk to prolong the QT interval for 7 days prior to starting study drug(s) or replaced by safe alternative medication.
  * Hypertension defined below:

Patients 1-12 years of age (pediatric) with blood pressure that is ≥ 95th percentile for age, height and gender at the time of enrollment

Patients who are ≥ 13 years of age (adolescents) with a blood pressure that is ≥130/80 mm of Hg at the time of enrollment.

* Note: If a BP reading prior to enrollment does not meet parameters, blood pressure should be rechecked and documented to be within eligibility range prior to patient enrollment.

* Inability to determine the QTc interval on the ECG (i.e.: unreadable or not interpretable) or QTc ≥ 450 msec as determined by screening ECG.
* Patient is currently receiving any of the following medications and cannot be discontinued 7 days prior to starting study drugs ribociclib and everolimus

  * Known strong inducers or inhibitors of CYP3A4/5, including grapefruit, grapefruit hybrids, pummelos, star-fruit, and Seville oranges
  * Strong and moderate inhibitors or inducers of CYP3A4/5
  * Substrates of CYP3A4/5 with a narrow therapeutic index
  * Other investigational and anti-neoplastic therapies, including chemotherapy, immunotherapy, target therapy, biological response modifiers
  * Medications that have a narrow therapeutic window and are predominantly metabolized through CYP3A4/5
  * Medications that have a known risk to prolong the QT interval or induce Torsades de Pointes
  * Herbal preparations/medications (except for vitamins) including, but not limited to: St. John's wort, Kava, ephedra (ma huang), gingko biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto, black cohosh and ginseng. Patients should stop using all herbal medications and dietary supplements at least 7 days prior to first dose of study treatment.
* Bleeding Disorder Patient is currently receiving warfarin or other coumadin-derived anticoagulant for treatment, prophylaxis or otherwise. Therapy with heparin, low molecular weight heparin (LMWH) or fondaparinux is allowed as long as patient has adequate coagulation defined as: aPTT INR≤1.5 x upper limit of normal.
* Patient has a history of non-compliance to medical regimen.
* Known need for major surgery within 14 days of the first dose of ribociclib and everolimus. Gastrostomy, insertion of a G tube, Ventriculo-peritoneal shunt, endoscopic ventriculostomy and central venous access are NOT considered major surgery.

Ages: 12 Months to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2017-11-14 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | 6 months
  Number of individual toxicities and incidence of significant delays
Estimate the maximum tolerated dose and/or recommended phase 2 dose of ribociclib combined with everolimus | 28 days
  number of dose limiting toxicities experienced at each dose level
Pharmacokinetics of combination of ribociclib and everolimus | 7 days
  Plasma concentration of ribociclib and everolimus over time

SECONDARY OUTCOMES:
Time from diagnosis to death - overall survival | 48 months
  Overall survival is defined as the time from diagnosis to death.
Number of patients with observed pseudoprogression | 12 months
  the assessment of true vs. pseudoprogression will be based on the tumor measurements from subsequent scans
Whole exome sequencing to explore biology of DIPG and HGG tumors | 24 months
  Genetic sequence analysis

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Levine Cancer Institute, Charlotte, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Texas Children's Hospital, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided
IPD would only be shared following publication of the study.